CLINICAL TRIAL: NCT01008917
Title: Phase I Trial of the Combination of Temsirolimus and Sorafenib in Advanced Hepatocellular Carcinoma
Brief Title: Temsirolimus and Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC# 09455; NCT01013519 (obsolete NCT alias)
Record Dates: First submitted 2009-10-30; First posted 2009-11-06 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; HCC; Liver cancer; Hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single treatment-non randomized study (Experimental): Phase I study is to test the safety of the combination of sorafenib with temsirolimus at different dose levels
  Interventions: Drug: sorafenib with temsirolimus

INTERVENTIONS:
Drug: sorafenib with temsirolimus — Weekly intravenous temsirolimus with daily oral sorafenib
  Other Names: Torisel; Nexavar

SUMMARY:
This is a Phase I study, which means that the goal is to see if the combination of Temsirolimus and Sorafenib is safe in patients with Hepatocellular Carcinoma. Sorafenib is a standard treatment for Hepatocellular Carcinoma. Temsirolimus is used to treat cancer in the kidneys. It is hoped that the addition of Temsirolimus will make Sorafenib more effective against Advanced Hepatocellular Carcinoma, however this can not be guaranteed. The addition of Temsirolimus to Sorafenib is not an FDA approved treatment for Advanced Hepatocellular cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a leading cause of cancer death worldwide with an incidence of over 600,000 new cases and almost as many deaths annually.1 Advanced stages of disease at diagnosis often preclude curative treatments, and the overall prognosis of patients diagnosed with advanced HCC remains dismal with median survival of approximately 8 months.2-4 Until recently, systemic therapies for advanced HCC have demonstrated minimal benefit in these patients, largely due to compromised hepatic function from underlying liver disease as well as intrinsic tumor chemoresistance.5-9 In the past year, however, publication of the Sorafenib Hepatocellular Carcinoma Assessment Randomized Protocol (SHARP) phase III trial demonstrated a significant improvement in overall survival (OS) in patients with advanced HCC treated with the biologic agent, sorafenib.4 Despite improvements in outcome with sorafenib, however, the median OS for patients with advanced HCC remains less than a year, and new therapies and combinations are in great need to combat this grim disease.

Sorafenib is a small molecule bi-aryl urea with multikinase inhibitor activity. A primary target is the serine-threonine kinase, Raf-1. Sorafenib also has antiangiogenic activity, inhibiting receptor tyrosine kinases including vascular endothelial growth factor (VEGF) receptors 2 and 3 and the platelet derived growth factor receptor (PDGFR).10-12 Preclinical studies in HCC show that Raf-1 kinase signaling along with prolific tumor angiogenesis are common features, providing a molecular rationale for the efficacy of this agent.11,13-16 Radiographically, HCC is a hypervascular tumor, providing additional clinical relevance to the exuberant angiogenesis observed in this tumor type in the preclinical setting.15 The efficacy of sorafenib in the SHARP trial validates the importance of these signaling pathways in HCC.

Another signaling pathway which may play a role in hepatocarcinogenesis is the phosphatase and tensin homolog (PTEN)/phosphatidylinositol-3'kinase (PI-3'K)/AKT pathway which activates the mammalian target of rapamycin (mTOR) kinase, in turn triggering multiple downstream cell growth, survival, and angiogenesis signals.26-28 Dysregulated phosphorylation and activation of mTOR signaling may occur due to loss of function of the PTEN tumor suppressor gene, constitutive activation of PI-3'K, or activation of AKT by aberrant upstream growth factor receptor signaling.27 Activated mTOR forms complexes with other proteins, including regulatory associated protein of mTOR (Raptor) and Rictor.26 The mTOR-Raptor complex in turn phosphorylates protein 70 S6 kinase (p70S6K) as well as eukaryotic initiation factor 4E (eIF-4E) binding protein-1 (4E-BP1). P70S6K and 4E-BP1 regulate translation of a host of proteins, including several proteins involved in cell proliferation. Signaling through mTOR also stimulates angiogenesis.26,28-30 Activation of mTOR may induce endothelial cell proliferation as well as increase levels of hypoxia inducible factor (HIF)-1α and HIF-2α, potentially via p70S6K-mediated translation versus decreased oxygen-dependent degradation.31-33 HIFs induce angiogenesis in response to cellular hypoxia by transcriptional activation of target genes including VEGF.32,34,35

The mTOR inhibitor, sirolimus, is a macrocyclic lactone rapamycin produced by the soil bacterium, Streptomyces hygroscopicus. Sirolimus demonstrates fungicidal, immunosuppressive, and antiproliferative properties and is widely used as an immunosuppressant in transplant patients to prevent allograft rejection.26,36 Inhibitors of mTOR are also under investigation as potential anti-cancer agents in multiple human malignancies due to the known proliferative effects of mTOR activation. Temsirolimus, everolimus, and deforolimus are derivatives of sirolimus with similar antiproliferative properties in vitro.26

Temsirolimus is a soluble ester analogue of sirolimus.37 Temsirolimus has been approved by the FDA for treatment of advanced renal cell carcinoma (RCC) and demonstrated a survival benefit as monotherapy by comparison with interferon alpha in a multicenter phase III trial.38,39 In that trial, 626 patients with previously untreated, poor prognosis, metastatic RCC were randomized to receive temsirolimus 25 mg intravenously weekly, 3 million units of interferon alpha subcutaneously three times weekly, or combination therapy with 15 mg of temsirolimus weekly plus 6 million units of interferon alpha three times weekly.39 The primary endpoint, overall survival, was 10.9 months in the temsirolimus group, by comparison with 7.3 months with interferon alpha and 8.4 months with combination therapy; both overall survival and progression free survival (PFS) were significantly prolonged in the temsirolimus group by comparison with interferon alpha alone (P = 0.008 and P < 0.001, respectively).

Combination of molecularly targeted therapies offers the theoretical potential for additive or synergistic inhibition of shared targets as well as targets in parallel pathways which may provide escape mechanisms from single-pathway inhibition. In the case of mTOR inhibitors, combination therapy with Ras pathway inhibition may augment efficacy by blocking a pathway upstream of mTOR kinase, while combination with antiangiogenic agents may enhance antiangiogenic effect.26,27

ELIGIBILITY:
Inclusion Criteria

* Histologically or clinically* diagnosed AJCC stage III or IV HCC not amenable to curative resection and with no prior systemic cytotoxic or molecularly-targeted therapies. *Clinical diagnosis is acceptable if tumor meets radiographic criteria.
* Age ≥ 18 years.
* Child-Pugh score A or score of B with 7 points only and bilirubin ≤ 2 mg/dL.
* ECOG performance status ≤ 2.
* Radiographically measurable disease in at least one site not previously treated with chemoembolization, radioembolization, or other local ablative procedures.
* Prior chemoembolization, local ablative therapies, or hepatic resection permitted if completed ≥ 6 weeks prior to study enrollment and if criterion 6 is present.
* Prior radiation for bone or brain metastases is permitted if patient is now asymptomatic and has completed all radiation and steroid therapy (if applicable) for brain or bone metastases ≥ 2 weeks prior to study enrollment.
* Treatment with appropriate antiviral therapy for patients with active HBV infection is required.
* Treatment for clinically-significant hyperglycemia, hyperlipidemia, or hypertension that develops on study is required.
* Baseline blood pressure must be adequately controlled with or without antihypertensive medications prior to enrollment (systolic < 140 mm Hg, diastolic < 90 mm Hg).
* Baseline cholesterol must be < 350 mg/dL and triglycerides < 300 mg/dL (with or without the use of antihyperlipidemic medications).
* Baseline fasting blood glucose must be ≤ 140 mg/dL and hemoglobin A1c less than 7% (with or without the use of anti-diabetic medications).
* Adequate baseline organ and marrow function as defined below:
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 75,000/mcL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 2 mg/dL or ≤ 1.5 times ULN
* AST(SGOT)/ALT(SGPT) ≤ 5 times ULN
* INR ≤ 1.5 times ULN
* Albumin ≥ 2.8 g/dL
* Creatinine ≤ 1.5 times ULN
* Able to tolerate oral therapy.
* Ability to give written informed consent and willingness to comply with the requirements of the protocol.
* Effective means of contraception are required in fertile, sexually-active patients.

Exclusion Criteria

* Mixed tumor histology or fibrolamellar variant tumors are excluded.
* Prior antiangiogenic therapy (including thalidomide, sorafenib, sunitinib, or bevacizumab).
* Prior treatment with mTOR inhibitor or other molecularly targeted therapy.
* Prior systemic cytotoxic therapies for HCC (chemoembolization is permitted if inclusion criteria are met).
* Treatment with other investigational agents.
* Immunosuppressive medications including systemic corticosteroids unless used for adrenal replacement, appetite stimulation, acute therapy for asthma or bronchitis exacerbation (≤ 2 weeks), or antiemesis.
* Patients with known HIV infection are excluded.
* Patients who have undergone liver transplantation are excluded.
* Symptomatic brain or bone metastases; prior radiation and/or steroid therapy for brain or bone metastases (if applicable) must be completed ≥ 2 weeks prior to study enrollment.
* History of seizure disorder requiring antiepileptic medication or brain metastases with seizures.
* Serious non-healing wound, ulcer, bone fracture, or abscess.
* Patients requiring chronic anticoagulation with warfarin are excluded. Patients treated with low molecular weight heparin or unfractionated heparin are eligible if on a stable dose without evidence of clinically significant bleeding for at least 2 weeks prior to enrollment.
* Active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ.
* Uncontrolled intercurrent illness.
* No required concomitant medications with potential for significant interaction with study drugs.
* Any other condition that compromises compliance with the objectives and procedures of this protocol, as judged by the Study Chair, is also grounds for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2012-09-12 (Actual); Study Completion 2013-06-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | up to 14 months after initial dose

SECONDARY OUTCOMES:
Determine safety/toxicity profile of temsirolimus in combination with sorafenib | Treatment Period up to 22 cycles estimated to be up to 88 weeks
  each cycle is 4 weeks long
Describe pharmacokinetics of temsirolimus alone in the cohort of 6 subjects treated at MTD | Three cycles of treatment estimated to be 12 weeks
  each cycle is 4 weeks long
Describe pharmacokinetics of temsirolimus in combination with sorafenib in the cohort of 6 subjects treated at MTD | Three cycles of treatment estimated to be 12 weeks
  each cycle is 4 weeks long
Incidence of progression-free survival, overall survival, and disease control rate | 4 weeks (± 5 days) after removal from study or until death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Robin K Kelley, MD, Principal Investigator — University of California, San Francisco; Alan P Venook, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois